CLINICAL TRIAL: NCT03693989
Title: Clinical Study of the Efficacy of the Ophthalmic Emulsion PRO-145 for the Management of Inflammation and Pain After Phacoemulsification Compared to Prednisolone Acetate 1%.
Brief Title: Clinical Study of the Efficacy of the Ophthalmic Emulsion PRO-145 for Inflammation and Pain After Phacoemulsification
Acronym: PRO-145/III
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Laboratorios Sophia S.A de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SOPH145-0716 / III
Record Dates: First submitted 2018-10-01; First posted 2018-10-03 (Actual); Results first posted 2019-12-02 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Cataract
Keywords: corticosteroid; anti-inflammatory steroid; phacoemulsification
MeSH Terms: conditions — Cataract | interventions — prednefrin; difluprednate

STUDY DESIGN:
Intervention Model Description: double-blind, controlled, parallel group, multicentre, randomized
Who Masked: Participant, Investigator
Masking Description: Blinding and masking The blinding will correspond to the research subject and the principal investigator. In addition, the statistical analysis will be carried out in a blinded manner in the case of a partial and final analysis.
  The masking will be carried out using boxes in the identical primary packaging in the two groups and re-labeling the bottles of both interventions.
  Blinding for the research subject and the researcher will be done by replacing the commercial labels in the case of the comparator in the bottles and the use of identical labels that contain the assignment number.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRO-145. (Experimental): Difluprednate 0.05%. Prepared by Sophia Laboratories, S.A. of C.V., Zapopan, Jalisco, Mexico.
  Interventions: Drug: Difluprednate 0.05%
- Prednefrin (Active Comparator): Prednefrin® SF. Prednisolone Acetate 1%. Prepared by Allergan, S.A. of C.V.
  Interventions: Drug: Prednefrin

INTERVENTIONS:
Drug: Difluprednate 0.05% — Dosage: 1 drop 4 times a day (every 4 hours) during the period of vigil in the operated eye, for 14 days. Dose reduction for 14 days at the discretion of the principal investigator.
  Other Names: PRO-145
  Arms: PRO-145.
Drug: Prednefrin — 1 drop 4 times a day (every 4 hours) during the period of vigil in the operated eye, for 14 days. Dose reduction for 14 days at the discretion of the principal investigator.
  - Route of administration: topical ophthalmic
  Other Names: Difluprednate
  Arms: Prednefrin

SUMMARY:
objective: To evaluate the efficacy of the ophthalmic emulsion PRO-145 in the treatment of inflammation and pain after phacoemulsification.

Hypothesis:

The use of the ophthalmic emulsion PRO-145 is effective in decreasing the inflammatory response evaluated by means of cellularity in the anterior chamber, after phacoemulsification.

Methodology:

Phase III clinical trial, double-blind, controlled, parallel group, multicentre, randomized.

Number of patients:

178 subjects divided into 2 groups (89 subjects per group), who will provide an eye for the evaluation of efficacy.

Diagnosis and main inclusion criteria:

Diagnosis: Postoperative phacoemulsification and foldable intraocular lens placement in a bag.

DETAILED DESCRIPTION:
The study subjects will be recruited from various research centers in western and central Mexico.

Each research center has a monitoring plan specified according to the recruitment capabilities of the same, which must be at least once a month, where the queries of your data entered into the electronic case report report will be reported to the center. (e-CRF) for which it has as time limit the next monitoring visit to make the pertinent changes.

The report of adverse events will be made according to the standard operating procedure (PNO) where it specifies, according to Official Mexican Standard 220 (NOM 220), that the signs or symptoms of adverse events will be reported based on the Medical Dictionary. for Regulatory Activities, for which the sponsor has version 20.1 in Spanish. For serious adverse events (SAEs) will be reported in accordance with the standardized operation procedure of pharmacovigilance of the sponsor, which adheres to the guidelines of NOM 220 and international regulations, these will be reported in the regulatory framework to the regulatory entity within a period of time no more than 7 days.

The study is registered in the National Registry of Clinical Trials (RNEC), entity equivalent to Clinical Trials in Mexico.

The quality assurance plan is carried out by the sponsor through the Quality Assurance agent in Clinical Research, whose function is to conduct inspections and audits of the research sites to document and generate reports of deviations from the protocol. In addition to the visits of the monitoring plan, the reliability of the data is guaranteed.

To verify the integrity, veracity and reliability of the data entered into the e-CRF, the monitors of each center will check the information uploaded to the portal with that reported in the source document of the principal investigator (PI), such as clinical notes, clinical history and documents. and formats attached to the research protocol, physical case report format, as well as those provided by the sponsor to the PI (subject's diary and quality and satisfaction survey).

The e-CRF used for this clinical study is provided by an internationally certified provider with the highest quality standards, protection of information under current regulations and confidentiality guarantee. The information that the PIs enter into the e-CRF is collated and verified by the clinical monitors and by the service provider's personnel, later reviewed and approved by the medical ophthalmologist researcher and by the Clinical Security Pharmacologist, who authorize the monitored data of clinical information and safety of the study molecule, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Age ≥ 18 years.
* Both sexes.
* Postoperative cataract surgery by phacoemulsification. o That they have met the criteria for phacoemulsification and a classification of the lens opacity classification system (LOCS) III cataract of Opalescence of the nucleus (NO) ≥2 and Kernel color (NC) ≥2.

Exclusion Criteria:

* Pregnant women, lactating or planning to get pregnant.
* Women of reproductive age and who do not have a hormonal contraceptive method, intrauterine device or bilateral tubal obstruction.
* Participation in another clinical research study ≤ 30 days before the baseline visit.
* Have previously participated in this same study with the contralateral eye.
* That they can not comply with their attendance at appointments or with all the requirements of the protocol.

Medical and therapeutic criteria.

* Surgery in both eyes in the same surgical shift.
* Time> 24 hours after having surgery.
* Intraocular lens placement outside the bag.
* Presentation of rupture of the posterior capsule, with or without the presence of vitreous.
* Carrying out an iridectomy, or lesion of the pupillary sphincter during phacoemulsification surgery.
* Scheduled for surgical intervention in the contralateral eye during the study period.
* History of glaucoma or ocular hypertension.
* History of increased Intraocular pressure (IOP) with the use of steroids.
* Intraocular pressure (IOP) ≥24.
* History of uveitis.
* Presence of corneal abrasion or corneal ulceration in the study eye.
* Use of steroids or topical non steroidal anti inflammatory drugs, 24 hours prior to surgery and until the start of instillation of investigational drugs.
* Use of anticoagulants, systemic steroids or immunomodulators in the last two weeks
* Periocular injection of any steroid in the study eye 4 weeks before the start of the instillation of the investigational drugs.
* Use of storage steroids 2 months prior to the start of instillation of investigational drugs.
* Presence or suspicion of keratitis and / or viral, bacterial or fungal conjunctivitis.
* Presence or suspicion of endophthalmitis.
* Presence or suspicion of toxic syndrome of the anterior segment.
* Severe corneal edema that does not allow assessment of the anterior chamber
* Macular diseases.
* Diabetes Mellitus with glycosylated hemoglobin (A1C) ≥ 6.5% (48 mmol / mol) or fasting glucose (no caloric intake by ≥ 8 hours) of ≥ 126 mg / dL (7.0 mmol / L).
* Any disease or condition that requires the use of topical or systemic nonsteroidal anti-inflammatories (NSAIDs) during the time of intervention.
* Any disease or condition that requires the use of steroids other than topical ophthalmic application.
* Subjects with a single eye.
* Any condition or disease that at the discretion of the principal investigator (IP) does not make the subject suitable for the study.
* Known hypersensitivity to the components of the products under investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2018-10-04 (Actual); Primary Completion 2019-08-07 (Actual); Study Completion 2019-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leopoldo Baiza Durán, MD, Study Director — Laboratorios Sophia S.A de C.V.
Locations (5):
- Mexico (5):
  - Catarata y Glaucoma de Occidente, Guadalajara, Jalisco
  - Novam y Vita, Guadalajara, Jalisco
  - Vision Cirugia Ambulatoria, Monterrey, Nuevo León
  - Hospital de la luz, Mexico City
  - Fundación de asistencia privada Conde de Valenciana, Mexico City

REFERENCES:
- [Derived] Palacio-Pastrana C, Chavez-Mondragon E, Soto-Gomez A, Suarez-Velasco R, Montes-Salcedo M, Fernandez de Ortega L, Nasser-Nasser L, Baiza-Duran L, Olvera-Montano O, Munoz-Villegas P. Difluprednate 0.05% versus Prednisolone Acetate Post-Phacoemulsification for Inflammation and Pain: An Efficacy and Safety Clinical Trial. Clin Ophthalmol. 2020 Jun 12;14:1581-1589. doi: 10.2147/OPTH.S254705. eCollection 2020. PMID 32606573

RESULTS

PARTICIPANT FLOW:
Groups:
- Prednefrin: Prednefrin® SF. Prednisolone Acetate 1%. Prepared by Allergan, S.A. of C.V.
  Prednefrin: 1 drop 4 times a day (every 4 hours) during the period of vigil in the operated eye, for 14 days. Dose reduction for 14 days at the discretion of the principal investigator.
  - Route of administration: topical ophthalmic
Period: Overall Study
Arm/Group | PRO-145. | Prednefrin
Started | 88 | 90
Completed | 85 | 86
Not Completed | 3 | 4
Not completed — Protocol Violation | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PRO-145. | Prednefrin | Total
Number analyzed (Participants) | 85 | 86 | 171
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.9 (11.6) | 64.7 (12.4) | 65.48 (11.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 49 | 93
  Male | 41 | 37 | 78
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 85 | 86 | 171
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Mexico | 85 | 86 | 171

OUTCOME MEASURES:

1. Primary Outcome: Visual Ability (VA)
Description: The VA will be evaluated basally, without refractive correction with the Snellen chart. Which will be located in a place with adequate lighting, natural or artificial and at a distance of 3 meters from the subject to be evaluated. The result of the Snellen fraction will be transformed to its decimal equivalent in LogMAR, ex. 20/20= 1.0, 20/25=0.8, 20/40= 0.5, 20/200= 1.0, etc. The subjects will be averaged by group.
Time Frame: day 28 at the final visit
Population: the analysis was performed per protocol (PP)
Measure: Mean (Standard Deviation); unit: units on a scale (LogMAR)
Arm/Group | PRO-145. | Prednefrin
Number analyzed (Participants) | 85 | 86
units on a scale (LogMAR) | 0.91 (0.1) | 0.87 (0.2)
Statistical Analysis 1: Comparison: PRO-145. vs Prednefrin; Test type: Other; p = 0.065, t-test, 2 sided; The study analysis was comparative, it was only sought to determine if the difference between treatments is statistically significant or not

2. Primary Outcome: Adverse Events
Description: The evaluation of adverse events requires a questioning conducted by the principal investigator and the appropriate exploratory techniques for its detection.
  the number of cases with adverse events will be reported per study arm
Time Frame: day 28 at the final visit
Population: The analysis of the study was per protocol
Measure: Number; unit: cases
Arm/Group | PRO-145. | Prednefrin
Number analyzed (Participants) | 85 | 86
cases | 93 | 89
Statistical Analysis 1: Comparison: PRO-145. vs Prednefrin; Test type: Other — The study analysis was comparative, it was only sought to determine if the difference between treatments is statistically significant or not; p = 0.223, t-test, 2 sided

3. Secondary Outcome: Cellularity in the Anterior Chamber
Description: unit: degrees, Direct observation (Biomicroscopy).
  Scale for anterior chamber cellularity. Grade/Number of cells
  Grade / Number of cells
  0 Any
  ½ + 1-5
  1. + 6-15
  2. + 16-25
  3. + 26-60
  4. + More than 60
  the cellularity will be measured according to the scale that is added next, considering as normal the degree 0, and abnormal any other degree.
Time Frame: day 28 at the final visit
Population: The analysis of the study was per protocol
Measure: Count of Participants; unit: Participants
Arm/Group | PRO-145. | Prednefrin
Number analyzed (Participants) | 85 | 86
Participants
  Grade 0 | 75 | 76
  Grade 1/2 | 8 | 6
  grade 1 | 2 | 4
  grade 2 | 0 | 0
  grade 3 | 0 | 0
  grade 4 | 0 | 0
Statistical Analysis 1: Comparison: PRO-145. vs Prednefrin; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.621, Chi-squared, Corrected

4. Secondary Outcome: Clinical Corneal Edema
Description: The evaluation of clinical edema will be evaluated by the Efron scale, which is a series of factorial sections of the cornea, including features such as grooves and folds. The Efron scale has a strong correlation with variations in intensity. The number will be reported according to the rating awarded.
  Efron Scale: 0 Normal, 1 very slight, 2 mild, 3 moderate and 4 severe.
Time Frame: day 28 at the final visit
Population: The study analysis was comparative, it was only sought to determine if the difference between treatments is statistically significant or not.
Measure: Count of Participants; unit: Participants
Arm/Group | PRO-145. | Prednefrin
Number analyzed (Participants) | 85 | 86
Participants
  Normal (0) | 85 | 83
  Very mild (1) | 0 | 3
  Mild (2) | 0 | 0
  Moderate (3) | 0 | 0
  Severe (4) | 0 | 0
Statistical Analysis 1: Comparison: PRO-145. vs Prednefrin; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.246, Fisher Exact

5. Secondary Outcome: Flare
Description: In the presence of intraocular inflammation, the increased permeability of the non-pigmented layer of the ciliary epithelium, the posterior epithelium of the iris and the vascular endothelium of the iris results in the accumulation of cells and proteins (visible to the examiner as flare) in the anterior chamber. Using a light beam of 0.2mm X 0.2mm directed obliquely to the anterior chamber with a forward inclination of the light source (slit lamp tower) the degree of flare and cellularity will be determined according to the group of work of standardization for the nomenclature of uveitis.
  Flare scale
  0 There is no flare
  1. + Mild
  2. + Moderate (iris and crystalline clearly visible)
  3. + Marking (iris and crystalline slightly blurred)
  4. + More than 60 (fibrin)
Time Frame: day 28 at the final visit
Measure: Count of Participants; unit: Participants
Arm/Group | PRO-145. | Prednefrin
Number analyzed (Participants) | 85 | 86
Participants
  0 | 84 | 86
  1+ | 1 | 0
  2+ | 0 | 0
  3+ | 0 | 0
  4+ | 0 | 0
Statistical Analysis 1: Comparison: PRO-145. vs Prednefrin; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.497, Fisher Exact

6. Secondary Outcome: Central Thickness of the Retina
Description: By means of optical coherence tomography (OCT) the Retinal central thickness (GCR) will be measured. OCT is a noninvasive imaging test that uses light waves to take photographs of the cross section of the retina (the light-sensitive tissue that lines the back of the eye).With a OCT, each of the characteristic layers of the retina can be observed, allowing mapping and measuring its thickness a micrometer result will be obtained and the analysis will be carried out between groups.
Time Frame: day 28 at the final visit
Population: The analysis of the study was per protocol
Measure: Mean (Standard Error); unit: microns
Arm/Group | PRO-145. | Prednefrin
Number analyzed (Participants) | 85 | 86
microns | 253.59 (26.9) | 263.38 (36.4)
Statistical Analysis 1: Comparison: PRO-145. vs Prednefrin; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.047, t-test, 2 sided

7. Secondary Outcome: Conjunctival Hyperemia
Description: Conjunctival hyperemia is defined as the simplest reaction of the conjunctiva to a stimulus, a red appearance secondary to the vasodilation of the conjunctival vessels of variable intensity, we will use the Efron scale for conjunctival hyperemia.
  0 normal
  1. very slight
  2. mild
  3. moderate
  4. severe
Time Frame: day 28 at the final visit
Population: The analysis of the study was per protocol
Measure: Count of Participants; unit: Participants
Arm/Group | PRO-145. | Prednefrin
Number analyzed (Participants) | 85 | 86
Participants
  Normal (0) | 78 | 73
  Very mild (1) | 5 | 11
  Mild (2) | 2 | 2
  Moderate (3) | 0 | 0
  Severe (4) | 0 | 0
Statistical Analysis 1: Comparison: PRO-145. vs Prednefrin; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.300, Chi-squared, Corrected

8. Secondary Outcome: Intraocular Pressure
Description: Tonometry is the objective measure of Intraocular pressure, based primarily on the force required to flatten the cornea, or the degree of corneal indentation produced by a fixed force. Goldman's tonometry is based on the Imbert-Fick principle. the result will be expressed in millimeters of mercury and the comparison between groups will be carried out
Time Frame: day 28 at the final visit
Population: The analysis of the study was per protocol
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | PRO-145. | Prednefrin
Number analyzed (Participants) | 85 | 86
mmHg | 13.88 (3.0) | 13.04 (2.4)
Statistical Analysis 1: Comparison: PRO-145. vs Prednefrin; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.045, t-test, 2 sided

9. Secondary Outcome: Symptomatology Post Instillation
Description: The subject will be questioned if after applying the medication he felt burning, pruritus, a foreign body sensation and blurred vision.
  Presence or absence: it will be marked as present (1) or absent (0) for each of the symptoms questioned
Time Frame: day 28 at the final visit
Population: The analysis of the study was per protocol
Measure: Count of Participants; unit: Participants
Arm/Group | PRO-145. | Prednefrin
Number analyzed (Participants) | 85 | 86
Participants
  burning eyes | 12 | 8
  itching eyes | 1 | 0
  foreign body sensation eyes | 0 | 2
  blurred vision | 2 | 3
Statistical Analysis 1: Comparison: PRO-145. vs Prednefrin; burning eyes comparison; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.346, Fisher Exact
Statistical Analysis 2: Comparison: PRO-145. vs Prednefrin; Itching eyes comparison; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.489, Fisher Exact
Statistical Analysis 3: Comparison: PRO-145. vs Prednefrin; foreign body sensation eyes comparison; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.497, Fisher Exact
Statistical Analysis 4: Comparison: PRO-145. vs Prednefrin; blurred vision comparison; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 1.000, Fisher Exact

ADVERSE EVENTS:
Time Frame: Adverse events were monitored throughout the study, for at least 10 months.
Arm/Group | PRO-145. | Prednefrin
All-Cause Mortality (participants affected / at risk) | 0/85 | 0/86
Serious Adverse Events (participants affected / at risk) | 1/85 | 0/86
Other Adverse Events (participants affected / at risk) | 55/85 | 45/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PRO-145. (N=85) | Prednefrin (N=86)
acute myocardial infarction (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PRO-145. (N=85) | Prednefrin (N=86)
ocular burning (Eye disorders) | 46 (46) | 35 (35)
blepharospasm (Eye disorders) | 0 (0) | 1 (1)
headache (Nervous system disorders) | 0 (0) | 3 (3)
anterior chamber cellularity (Eye disorders) | 0 (0) | 1 (1)
infectious conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
flu (Infections and infestations) | 0 (0) | 2 (2)
stomach ache (Gastrointestinal disorders) | 0 (0) | 1 (1)
ocular pain (Eye disorders) | 2 (2) | 2 (2)
chemosis (Eye disorders) | 0 (0) | 1 (1)
Diabetic Macular Edema (Eye disorders) | 0 (0) | 1 (1)
pharyngotonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 3 (3) | 3 (3)
ocular hypertension (Eye disorders) | 2 (2) | 0 (0)
urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
eyelid inflammation (Eye disorders) | 0 (0) | 1 (1)
tearing (Eye disorders) | 1 (1) | 0 (0)
neovascular macular membrane (Eye disorders) | 0 (0) | 1 (1)
myodesopsia (Eye disorders) | 1 (1) | 1 (1)
red eye (Eye disorders) | 3 (3) | 6 (6)
earache (Ear and labyrinth disorders) | 0 (0) | 1 (1)
paresthesia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
eye itching (Eye disorders) | 7 (7) | 6 (6)
rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
eye foreign body sensation (Eye disorders) | 15 (15) | 11 (11)
Irvine-Gass syndrome (Eye disorders) | 0 (0) | 1 (1)
head trauma (General disorders) | 1 (1) | 0 (0)
Blurred Vision (Eye disorders) | 9 (9) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-08): https://cdn.clinicaltrials.gov/large-docs/89/NCT03693989/Prot_SAP_000.pdf